CLINICAL TRIAL: NCT01171300
Title: Assessment of Response Before, During and After Neoadjuvant Chemoradiotherapy in Rectal Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S52399
Record Dates: First submitted 2010-07-13; First posted 2010-07-28 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Adenocarcinoma; Rectal Neoplasms
Keywords: staged T3-4 N0 and T1-4N1-2; adenocarcinoma of the rectum; rectum
MeSH Terms: conditions — Adenocarcinoma; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: 18F- FDG PET scans — We aim to investigate the value of FGD-PET for evaluating response before surgery. To achieve this, the patients will undergo 3 FDG-PET scans (at moment of diagnosis (staging), during chemoradiation (early response), 1-2 weeks before surgery (restaging))
Other: DW-MRI scans — We aim to investigate the value of DW-MRI for evaluating response before surgery. To achieve this, the patients will undergo 3 FDG-PET scans (at moment of diagnosis (staging), during chemoradiation (early response), 1-2 weeks before surgery (restaging))

SUMMARY:
Rectal cancer is a frequent but curable malignancy in the Western world. The golden standard in treating these patients consists of neoadjuvant chemoradiotherapy (CRT) followed by extensive surgery regardless of tumor response. The main question is whether extensive surgery can be avoided holding in mind that already a significant amount of patients reach a pathological complete response after radiochemotherapy. The goal of this study is dual. First of all, the investigators want to investigate the value of DW-MRI and 18FDG-PET in the assessment of response after neoadjuvant CRT in 100 patients with rectal cancer, to select those patients eligible for less invasive surgery. In the same patient group, the investigators will examine the biomarker potential of molecular characteristics of the tumor in blood and tissue. Using both molecular and radiological findings, the investigators want to predict pathological response after chemoradiotherapy and to select patients who may benefit from treatment adjustments during chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age.
* Patient's body weight is ≤ 120 kg.
* Histologically proven and evaluable (according to RECIST criteria) adenocarcinoma of the rectum (tumour <15 cm from the anal verge), staged T3-4 N0 and T1-4N1-2.
* WHO PS ≤ 2
* Adequate bone marrow, hepatic and renal function (assessed within 14 days prior to study entry):
* Hemoglobin >10.0 g/dL,
* Absolute neutrophil count > 1.5 x 109/L,
* Platelet count > 100 x 109/L,
* Presence of adequate contraception in fertile patients. Adequate methods of contraception are: intra-uterine device, hormonal contraception, condom use with spermicide.
* Written informed consent must be given according to ICH/GCP and national/local regulations.

Exclusion Criteria:

* Evidence of distant metastases.
* Prior chemotherapy or radiotherapy for rectal cancer.
* Pregnant or breastfeeding women.
* Significant impairment of intestinal resorption (e.g. chronic diarrhea, inflammatory bowel disease).
* Known allergies to intravenous contrast agents.
* Contra-indications for magnetic resonance imaging (metal implants, claustrophobia, etc. ).
* Previous or concurrent malignancies at other sites with the exception of surgically cured or adequately treated carcinoma in-situ of the cervix and non-melanoma skin cancer.
* History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant precluding informed consent or interfering with compliance for oral drug intake.
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2010-10; Primary Completion 2015-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (ypT0N0) rate | 6-8 weeks after the end of chemoradiotherapy

SECONDARY OUTCOMES:
Pathologic downstaging (ypT0-2N0) rate and Tumour Regression Grade (TRG); according to Dworak et al. Response rate at time of surgery (RECIST criteria based on MRI); | 6-8 weeks after the end of chemoradiotherapy
Quality of mesorectal excision. | 6-8 weeks after the end of chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Karin Haustermans, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Gasthuisberg, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- See also: Related Info — http://www.uzleuven.be